CLINICAL TRIAL: NCT01577043
Title: Efficacy of Racecadotril in the Management of Acute Watery Diarrhea in Children
Brief Title: Efficacy of Racecadotril in Acute Watery Diarrhea in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Pediatrico Albina de Patino (Other)
Responsible Party: Principal Investigator, Giuseppe Grandy, Medical Chief of Nutrition Center, Centro Pediatrico Albina de Patino
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: protracec2011
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2011-06

CONDITIONS: Acute Diarrhea; Acute Gastroenteritis
Keywords: acute diarrhea; Racecadotril; children
MeSH Terms: interventions — racecadotril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Racecadotril (Active Comparator): intestinal antisecretory
  Interventions: Drug: Racecadotril
- cornstach solution (Placebo Comparator): Cornstarch powder diluted in distilled water
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Racecadotril — Racecadotril, 30 mg per sachet, dosage 1.5 mg./kg./day
  Other Names: Hidrasec
  Arms: Racecadotril
Other: Placebo — cornstarch powder diluted in distilled water, dosage 2.5 ml per dose
  Arms: cornstach solution

SUMMARY:
The purpose of this study is to determine the effect of racecadotril in acute watery diarrhea in children. The investigators will evaluate the effect of product versus placebo.

DETAILED DESCRIPTION:
Background: Treatment of acute diarrhea is based on the following various oral rehydration management guidelines. Lately other drugs currently under investigation as antisecretory drugs to shorten the diarrheal episode and can be used safely in children.

Objectives: To evaluate the effect of racecadotril in the treatment of children under 5 years of age with acute diarrhea.

Methods: A randomized clinical trial, controlled, double-blind. The investigators will have two groups of patients: One group will receive racecadotril plus oral rehydration and the other one will receive placebo plus oral rehydration; the parameters of evaluation are going to be the duration of diarrheal episode, number of stools by day, weight of stool, nutritional state.

ELIGIBILITY:
Inclusion Criteria:

* Acute watery diarrhea

Exclusion Criteria:

* Severe malnourishment
* Severe dehydration
* Systemic infections
* Coinfections

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Duration of diarrheal episode | five days
  Duration of diarrheal episode, time in which the watery stools will be normalized, an expected average of 5 days

SECONDARY OUTCOMES:
Duration of hospitalization | five days
  Participants was followed for the duration of hospitalization, we expected average of 5 days
Weight of stool | five days
  We expected the weight of the stool will diminish by about 5 days
Frequency of stool per day | five days
  We expected the frequency of stool will diminish by about 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Grandy, MD MSc, Study Director — Centro Pediatrico Albina de Ptino; Richard Soria, MD, Principal Investigator — Centro Pediatrico Albina de Patino; Jackeline Torrez, MD, Study Chair — Centro Pediatrico Albina de Patino
Locations (1):
- Centro Pediatrico Albina de Patino, Cochabamba, Departamento de Cochabamba, Bolivia